CLINICAL TRIAL: NCT07393815
Title: Physiological Responses to Graded Manual Pressure in Healthy Adults: a Randomized Experimental Study on Autonomic, Hormonal, Sensory and Vascular Outcomes
Brief Title: "Physiological Responses to Manual Pressure in Healthy Adults"
Acronym: VALIRAT1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VALIRAT 1
Record Dates: First submitted 2025-12-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
Keywords: Autonomic Nervous System; Manual Therapy; Pain
MeSH Terms: conditions — Pain | interventions — Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Sustained Pressure (Experimental): Participants receive a graded manual pressure protocol applied as sustained pressure at a single point over the upper trapezius muscle (0, 25, 50, 75 and 90% of individual PPT, 2 minutes each level, randomized order).
  Interventions: Other: Graded Sustained Pressure
- Experimental: Longitudinal Kneading (Experimental): Participants receive the same graded pressure protocol applied as longitudinal kneading over a defined area of the upper trapezius muscle (0, 25, 50, 75 and 90% of individual PPT, 2 minutes each level, randomized order).
  Interventions: Other: "Manual Pressure Protocol"
- Experimental: Manual Therapy Protocols (Experimental): Participants receive three standardized manual therapy protocols with increasing pressure in three separate sessions, with randomized order: (1) manual lymphatic drainage (~40 mmHg, approximately 40 minutes), (2) light-pressure massage (0.5-0.8 N/cm², 20-30 minutes) and (3) moderate-pressure massage (2-3 N/cm², 20 minutes), targeting the upper trapezius and related regions.
  Interventions: Other: Manual Therapy Protocols (DLM, light and moderate-pressure massage)

INTERVENTIONS:
Other: "Manual Pressure Protocol" — Manual pressure is applied over the upper trapezius muscle using five individualized pressure levels (0, 25, 50, 75 and 90% of the pressure pain threshold). Each level is applied for 2 minutes in a single experimental session, with randomized order and rest periods between applications. In the Sustained Pressure arm, pressure is maintained at a single point. In the Longitudinal Kneading arm, the same pressure levels are distributed along a predefined area using a kneading technique.
  Arms: Experimental: Longitudinal Kneading
Other: Manual Therapy Protocols (DLM, light and moderate-pressure massage) — Three standardized manual therapy protocols targeting the upper trapezius and related regions are applied in separate sessions with at least one day between them and randomized order: (1) manual lymphatic drainage (approx. 40 minutes at ~40 mmHg), (2) light-pressure massage (0.5-0.8 N/cm², 20-30 minutes) and (3) moderate-pressure massage (2-3 N/cm², 20 minutes). Pressure is monitored continuously with a hand-worn pressure sensor.
  Arms: Experimental: Manual Therapy Protocols
Other: Graded Sustained Pressure — Manual pressure applied over the upper trapezius using five individualized pressure levels (0, 25, 50, 75 and 95% of the pressure pain threshold) delivered as sustained pressure at a single point, 2 minutes per level in a single session, with randomized order and rest periods between applications.
  Arms: Experimental: Sustained Pressure

SUMMARY:
This randomized experimental study will investigate how different intensities and application patterns of manual pressure applied to the upper trapezius muscle affect physiological responses in healthy adults. Participants will be randomly assigned to one of three groups: (A) graded sustained pressure at a single point over the upper trapezius, (B) graded longitudinal kneading over a defined area of the upper trapezius, or (C) three standardized manual therapy protocols with increasing pressure (manual lymphatic drainage, light-pressure massage and moderate-pressure massage).

In groups A and B, five individualized pressure levels (0, 25, 50, 75 and 95% of each participant's pressure pain threshold) will be delivered for 2 minutes each in a single session. In group C, each participant will receive the three manual therapy protocols in separate randomized sessions. Autonomic (heart rate and heart rate variability), hormonal (capillary cortisol and VEGF in group C), sensory (mechanical pain thresholds), hemodynamic (blood pressure) and, in group C, vascular (left common carotid artery ultrasound) responses will be recorded before and after the interventions. The study will provide dose-response and mechanistic information to inform safer and more individualized manual therapy protocols.

DETAILED DESCRIPTION:
This prospective randomized experimental study will be conducted in healthy adults to characterize acute physiological responses to different intensities and patterns of manual pressure applied to the upper trapezius muscle. Participants will be randomly allocated to one of three experimental groups:

* Group A - Graded sustained pressure: a personalized pressure scale is defined based on the individual pressure pain threshold (PPT) measured with an algometer. Five pressure levels are set at 0% (contact without pressure), 25%, 50%, 75% and 95% of PPT, and applied as sustained pressure at a single point over the upper trapezius.
* Group B - Graded longitudinal kneading: the same personalized pressure scale (0, 25, 50, 75 and 95% of PPT) is applied as longitudinal kneading distributed over a predefined area of the upper trapezius.
* Group C - Manual therapy protocols: each participant receives three standardized manual therapy protocols in separate sessions, with randomized order: manual lymphatic drainage (approx. 40 minutes at ~40 mmHg), light-pressure massage (0.5-0.8 N/cm², 20-30 minutes) and moderate-pressure massage (2-3 N/cm², 20 minutes), all targeting the upper trapezius and related regions.

In groups A and B, the five pressure levels are each applied for 2 minutes in a single experimental session, in randomized order, with rest periods of at least 5 minutes between levels (extended if needed until heart rate returns within ±10% of baseline). In group C, each manual therapy protocol is applied in a separate session with at least one day between sessions. In all groups, heart rate and heart rate variability are recorded continuously with a chest strap, and skin temperature and skin conductance are continuously monitored with surface sensors. Blood pressure, mechanical pain thresholds (von Frey filaments at predefined trapezius and forearm sites), and capillary blood samples for cortisol are obtained at baseline and immediately after each pressure level or massage protocol. In group C, VEGF is also measured in capillary blood.

In group C only, duplex ultrasound of the left common carotid artery is performed under standardized conditions (semi-recumbent position, head rotated 45° to the right) before the manual therapy protocol and 10 minutes after its completion, to assess luminal diameter, intima-media thickness and peak systolic velocity. All pressure applications in all groups are monitored with a pressure-sensing system (Loadpad) placed on the therapist's hand.

A separate visit includes whole-body dual-energy X-ray absorptiometry (DEXA) to characterize body composition (total and segmental lean mass and fat mass). The main outcome is a heart rate variability index (e.g., RMSSD), while hormonal (cortisol, VEGF in group C), sensory (pain thresholds), hemodynamic (blood pressure) and vascular (carotid ultrasound in group C) measures are considered secondary outcomes. The study is powered assuming a large effect size on HRV based on previous massage research, with a planned sample size of 30 participants per group (N = 90).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Healthy volunteers without diagnosed cardiovascular, neurological or severe musculoskeletal disorders.
* No significant pain or pathology in the cervical, shoulder or upper back region that would interfere with pressure application.
* Ability to understand the study procedures and to provide written informed consent.
* Availability to attend the experimental session and the DEXA visit.

Exclusion Criteria:

* History of major cardiovascular disease (e.g., ischemic heart disease, heart failure, clinically significant arrhythmias, uncontrolled hypertension, stroke or transient ischemic attack).
* Neurological disorders affecting pain perception or autonomic function.
* Acute or chronic musculoskeletal conditions in the cervical or shoulder region that contraindicate manual pressure on the upper trapezius.
* Coagulation disorders or high-dose anticoagulant/antiplatelet therapy that increases bleeding risk.
* Dermatologic conditions or skin lesions at sensor placement or pressure application sites.
* Pregnancy or suspected pregnancy (due to DEXA scan).
* Regular use of medications with a major impact on autonomic or cardiovascular responses (e.g., beta-blockers, antiarrhythmics) that cannot be paused according to medical judgement.
* Substance abuse or acute alcohol/drug intake in the 24 hours prior to the experimental session.
* Any other condition that, in the opinion of the investigators, may compromise safety or compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) index | Baseline and after10 min
  Heart rate variability (HRV) will be recorded continuously using a chest strap. An HRV index (e.g., RMSSD or SDNN) will be calculated for predefined periods (baseline, during and after each pressure condition). The primary outcome will be the change in HRV across pressure levels and between intervention groups.

SECONDARY OUTCOMES:
Change in capillary cortisol level | Baseline and after10 min
  Capillary blood cortisol measured by ELISA; changes relative to baseline will be compared across pressure levels and groups.
Change in mechanical pain threshold (von Frey) | Baseline and after10 min
  Mechanical pain thresholds assessed with von Frey filaments at predefined sites (upper trapezius and forearm); changes across pressure levels and groups.
Change in blood pressure | Baseline and after10 min
  Systolic and diastolic blood pressure measured with a manual sphygmomanometer.
Change in skin temperature | Periprocedural
  Continuous recording throughout the session.
Change in skin conductance | Periprocedural
  Skin conductance (electrodermal activity) recorded as an index of sympathetic arousal.
Change in common carotid artery diameter | Baseline and after10 min
  Left common carotid artery luminal diameter (intima-intima) assessed by B-mode ultrasound; absolute and relative changes pre-post session. (Group C only)
Change in common carotid artery intima-media thickness (IMT) | Baseline and after10 min
  Left common carotid artery luminal diameter, intima-media thickness assessed by B-mode and Doppler ultrasound in group C before and 10 minutes after each manual therapy protocol.
Change in common carotid artery peak systolic velocity (PSV) | Baseline and after10 min
  Peak systolic velocity assessed by B-mode and Doppler ultrasound in group C before and 10 minutes after each manual therapy protocol.
Body composition (DEXA) | Baseline
  Total and segmental lean mass and fat mass, used as descriptive and potential modulators.
Change in capillary VEGF level | Baseline and after10 min
  Capillary blood VEGF (vascular endothelial growth factor) measured by ELISA in group C participants at baseline and immediately after each manual therapy protocol; changes relative to baseline will be compared across the three protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Unalmis Y, Muniroglu S (2026). Efficacy of fascial manipulation in musculoskeletal pain management: a decade in review (2015-2025). J. Bodyw. Mov. Ther. 46:147-156.
- [Background] Roura S, Álvarez G, Solà I, Cerritelli F (2021) Do manual therapies have a specific autonomic effect? An overview of systematic reviews. PLoS ONE 16(12): e0260642
- [Background] Picchiottino M, Leboeuf-Yde C, Gagey O, Hallman DM. (2019) The acute effects of joint manipulative techniques on markers of autonomic nervous system activity: a systematic review and meta-analysis of randomized sham-controlled trials. Chiropr Man Therap. 27:17.
- [Background] Petrova TV, Koh GY (2023). The Emerging Importance of Lymphatics in Health and Disease. J. Clin. Invest. 133(12):e171582
- [Background] Pérez García R, Ruiz Miñarro R, Robledo Do Nascimento Y (2018) Efectos del DLM en la respuesta inmunitaria específica. Congreso Internacional de Fisioterapia 1:1
- [Background] Mínguez-Esteban, I., De la Cueva-Reguera, M., Abuín-Porras, V., Romero-Morales, C., Almazán-Polo, J., & Bravo-Aguilar, M. (2025). Acute sonographic changes in common carotid artery after NESA neuromodulation intervention in healthy adults: A randomized controlled clinical trial. Frontiers in Neuroscience, 19, 1526236
- [Background] • Lima CR, Fernandes Martins D, Reed WR (2020). Physiological responses induced by manual therapy in animal models: a scoping review. Front. Neurosci. 14:430
- [Background] Huggenberger R, Detmar M (2013). Lymphatic Function and Immune Regulation in Health and Disease. Lymph. Res. Biol. 11(1):1-17
- [Background] Diego MA, Field T (2009). Moderate pressure massage elicits a parasympathetic nervous system response. Int. J. Neurosci. 119:630-638
- [Background] Amoroso Borges BL, Bortolazzo GL, Neto HP. (2018) Effects of spinal manipulation and myofascial techniques on heart rate variability: A systematic review. J Bodyw Mov Ther. 22:203-208
- [Background] Alnefaie HA, Alserahi YS, Kattan MI, Alsaedi SS, Shafei SI, Alotaibi AA, Alfahemy MM, Alqethmi FS, Alkhattabi AH (2025). Physiotherapy in the management of musculoskeletal disorders: a systematic review. The review of diabetic studies 21:102-114.